CLINICAL TRIAL: NCT00157157
Title: Recombinant Antihemophilic Factor Manufactured and Formulated Without Added Human or Animal Proteins (rAHF-PFM): Evaluation of Immunogenicity, Efficacy, and Safety in Previously Untreated Patients With Hemophilia A
Brief Title: Efficacy and Safety Study of a Recombinant Protein-Free Manufactured Factor VIII (rAHF-PFM) in Previously Untreated Hemophilia A Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060103; 2004-001623-38 (EudraCT Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
Keywords: Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm - All Participants (Experimental): All subjects enrolled in the study who meet the eligibility criteria.
  Interventions: Biological: Recombinant Antihemophilic Factor Manufactured and Formulated without Added Human or Animal Proteins (rAHF-PFM)

INTERVENTIONS:
Biological: Recombinant Antihemophilic Factor Manufactured and Formulated without Added Human or Animal Proteins (rAHF-PFM) — Treatment regimens were determined by the investigator, and may have been any combination of standard prophylaxis (25 to 50 IU/kg body weight, 3 to 4 times per week), investigator-determined prophylaxis, and/or on-demand treatment (dose selected by investigator).
  The treatment of bleeding episodes and perioperative management was at the discretion of the investigator and consistent with the institution's standard of care.
  For incremental recovery assessments, a single infusion at 50 +/- 5 IU/kg was to be given.
  Immune tolerance induction (ITI) therapy for subjects who developed factor VIII inhibitors was at the discretion of the investigator, based on the institution's guidelines or described in peer-reviewed literature, and was to be approved by the sponsor's medical director.
  rAHF-PFM was to be administered intravenously via bolus infusion, except for perioperative management when it may have been given either by continuous or bolus infusion.

SUMMARY:
The purpose of this study is to evaluate whether Antihemophilic factor, recombinant, manufactured protein-free (rAHF-PFM) is effective and safe in the treatment of hemophilia A patients who have not been treated with factor VIII (FVIII) before.

ELIGIBILITY:
Inclusion Criteria:

* The subject has severe or moderately severe hemophilia A as defined by a baseline factor VIII level <= 2% of normal, as documented at screening
* The subject is < 6 years of age
* The subject's legally authorized representative has provided written informed consent

Exclusion Criteria:

* The subject has a history of exposure to factor VIII other than rAHF PFM or more than 3 infusions of commercially available rAHF PFM (i.e., ADVATE) within 28 days prior to screening, as determined by the subject's medical history. Any infusion of factor VIII replacement products prior to the 28-day period excludes the subject from participation
* The subject has received more than 3 infusions of rAHF PFM (commercially available and/or study product) between screening and prior to the initial recovery infusion
* The subject has a detectable inhibitor to factor VIII, as measured in the screening sample by the Nijmegen assay in the central laboratory
* The subject has a history of inhibitor to factor VIII at any time prior to screening
* The subject has a known hypersensitivity to rAHF PFM
* The subject has any 1 of the following laboratory abnormalities at the time of screening:

  1. Platelet count < 100,000/mm^3
  2. Hemoglobin concentration < 10 g/dL (100 g/L)
  3. Serum creatinine > 1.5 times the upper limit of normal (ULN) for age
  4. Total bilirubin > 2 times the ULN for age
* The subject has an inherited or acquired hemostatic defect other than hemophilia A (e.g., qualitative platelet defect or von Willebrand's disease)
* The subject is known to be seropositive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV), as determined by the subject's medical history
* At the time of enrollment, the subject has a clinically significant chronic disease other than hemophilia A
* The subject is currently participating in another investigational drug study, or has participated in any clinical study involving an investigational drug within 120 days of the screening visit
* The subject (or the subject's legally authorized representative) is identified by the investigator as being unable or unwilling to cooperate with study procedures
* The subject has received any blood product, including packed red blood cells (RBC), platelets, plasma, or cryoprecipitate

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2009-09-11 (Actual); Study Completion 2009-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (35):
- United States (17):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - New Hyde Park, New York
  - New York, New York
  - Philadelphia, Pennsylvania
  - Houston, Texas
- Vienna, Austria
- Toronto, Ontario, Canada
- France (6):
  - Caen
  - Le Kremlin-Bicêtre
  - Lyon
  - Marseille
  - Nantes
  - Paris
- Germany (4):
  - Bremen
  - Frankfurt
  - Hanover
  - Münster
- Milan, Italy
- San Juan, Puerto Rico
- Barcelona, Spain
- Stockholm, Sweden
- United Kingdom (2):
  - Cardiff, Wales
  - London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Ewenstein B., Patrone L, Schroth P, Spotts G, Fritsch S, Pavlova B, Ehrlich H. Efficacy of antihemophilic factor (recombinant), plasma/albumin-free method (rAHF-PFM) in bleed prevention. J Thromb Haemost. 2007; 5(Suppl 2): P-S-179.
- [Result] Ewenstein B., Patrone L, Schroth P, Spotts G, Fritsch S, Pavlova B, Ehrlich H. Efficacy of antihemophilic factor (recombinant), plasma/albumin-free method (rAHF-PFM) in bleed treatment. J Thromb Haemost. 2007; 5(Suppl 2)v: P-S-180.
- [Result] Shapiro A, Gruppo R, Pabinger I, Collins PW, Hay CR, Schroth P, Casey K, Patrone L, Ehrlich H, Ewenstein BM. Integrated analysis of safety and efficacy of a plasma- and albumin-free recombinant factor VIII (rAHF-PFM) from six clinical studies in patients with hemophilia A. Expert Opin Biol Ther. 2009 Mar;9(3):273-83. doi: 10.1517/14712590902729392. PMID 19216617
- [Derived] Auerswald G, Thompson AA, Recht M, Brown D, Liesner R, Guzman-Becerra N, Dyck-Jones J, Ewenstein B, Abbuehl B. Experience of Advate rAHF-PFM in previously untreated patients and minimally treated patients with haemophilia A. Thromb Haemost. 2012 Jun;107(6):1072-82. doi: 10.1160/TH11-09-0642. Epub 2012 Apr 4. PMID 22476554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the U.S., Canada, and Europe at 24 study sites.
Pre-assignment Details: Participants screened for maximum 21 days. Study was not randomized; it was an open-label evaluation. Prior to initial infusion, a minimum washout period of 3 days was required. 11 participants who enrolled did not receive any rAHF-PFM infusions (3 withdrew consent, 6 screen failures, 1 non-compliance with screening, 1 pre-existing low hemoglobin)
Groups:
- Previously Untreated Patients (PUPs): rAHF-PFM was dosed according to a therapeutic regimen which was determined by the investigator (ie: standard regimen [25 to 50 IU/kg body weight, 3 to 4 times per week]; a modified prophylactic regimen [dose and frequency selected by investigator] or on-demand treatment [dose selected by investigator]). The dosing regimen used to treat bleeding episodes (BEs) was at the discretion of the investigator and in accordance with the institution's standard of care for the type of bleeding episodes diagnosed.
Period: Overall Study
Arm/Group | Previously Untreated Patients (PUPs)
Started | 55
Completed | 44
Not Completed | 11
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Enrolled in another study | 1
Not completed — Met exclusion criteria | 1
Not completed — Inclusion not met- baseline FVIII value | 1

BASELINE CHARACTERISTICS:
Arm/Group | PUPs
Number analyzed (Participants) | 55
Age, Customized [Count of Participants; unit: Participants]
  <6 months | 21
  6-12 months | 26
  ≥13 months | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Factor VIII Inhibitor Development
Description: Percentage of treated participants who developed factor VIII inhibitors
Time Frame: Assessed during study period which was to be at least 75 exposure days or 3 years (whichever came first)
Population: Participants who received at least 1 infusion of rAHF-PFM
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | PUPs
Number analyzed (Participants) | 55
percentage | 29.1 [17.1 to 41.1]

2. Secondary Outcome: Bleeding Episodes Treated With 1 to ≥4 Infusions
Description: The number of bleeding episodes treated with 1, 2, 3, or ≥4 infusions of rAHF-PFM to achieve adequate hemostasis
Time Frame: Reported during study period which was to be at least 75 exposure days or 3 years (whichever came first)
Population: Participants who received at least 1 infusion of rAHF-PFM for the treatment of bleeding episodes
Measure: Number; unit: Bleeding episodes
Arm/Group | PUPs
Number analyzed (Participants) | 44
Bleeding episodes
  1 infusion | 356
  2 infusions | 107
  3 infusions | 35
  4 or more infusions | 19

3. Secondary Outcome: Assessment of Hemostasis for Treatment of Bleeding Episodes
Description: Number of rAHF-PFM-treated bleeding episodes with treater assessment of hemostasis (4-point ordinal scale): Excellent: Full pain relief & bleeding cessation within ~8 hrs of 1 infusion. Additional infusions may have been given to maintain hemostasis; Good: Definite pain relief and/or improvement in bleeding within ~8 hrs after infusion. Possibly requires >1 infusion for complete resolution; Fair: Probable or slight relief of pain & slight improvement in bleeding within ~8 hrs after infusion. Requires >1 infusion for complete resolution; or None: No improvement or condition worsens.
Time Frame: Reported during study period which was to be at least 75 exposure days or 3 years (whichever came first)
Population: Participants who received at least 1 infusion of rAHF-PFM and had at least 1 treated bleeding episode. The 1 rating of "none" was for the first 2 infusions, the last infusion was rated as "good".
Measure: Number; unit: bleeding episodes
Arm/Group | PUPs
Number analyzed (Participants) | 44
bleeding episodes
  Excellent | 258
  Good | 177
  Fair | 30
  None | 1
  Unknown/not assessed | 51

4. Secondary Outcome: Annualized Rate of Bleeding Episodes
Description: Number of bleeding episodes per subject annualized over 1 year for all etiologies
Time Frame: Reported during study period which was to be at least 75 exposure days or 3 years (whichever came first)
Population: Participants treated for at least 3 months with investigator-defined on-demand treatment (for dose) or prophylaxis (for dose and infusion frequency) for >80% of the treatment period
Measure: Median (Full Range); unit: bleeding episodes per subject per year
Arm/Group | PUPs
Number analyzed (Participants) | 43
bleeding episodes per subject per year | 4.95 [1.01 to 32.70]

5. Secondary Outcome: Weekly rAHF-PFM Utilization
Description: Weight-Adjusted Weekly Dose for Prophylaxis, On-Demand Treatment, and Perioperative Management. rAHF-PFM dose determined by the investigator (ie: standard regimen [25-50 IU/kg body weight, 3-4 times per week]; modified prophylactic regimen [dose and frequency selected by investigator] or on-demand treatment [dose selected by investigator]). Dosing to treat BEs was at investigator's discretion and in accordance with institution's standard of care. rAHF-PFM was administered I.V. via bolus infusion, except for perioperative management when it was given either by continuous or bolus infusion.
Time Frame: Reported during study period which was to be at least 75 exposure days or 3 years (whichever came first)
Population: as for outcome 4
Measure: Median (Full Range); unit: IU/kg
Groups:
- PUPs -During Prophylaxis: rAHF-PFM was dosed according to a therapeutic regimen which was determined by the investigator (ie: standard regimen [25 to 50 IU/kg body weight, 3 to 4 times per week]; a modified prophylactic regimen [dose and frequency selected by investigator]. The dosing regimen used to treat BEs was at the discretion of the investigator and in accordance with the institution's standard of care for the type of bleeding episode (BE) diagnosed.
- PUPs -During On-Demand Treatment: The dosing regimen used to treat BEs was at the discretion of the investigator and in accordance with the institution's standard of care for the type of BE diagnosed.
- PUPs -During Perioperative Management: rAHF-PFM was administered intravenously via bolus infusion, or continuous infusion. The dosing regimen used was at the discretion of the investigator and in accordance with the institution's standard of care.
Arm/Group | PUPs -During Prophylaxis | PUPs -During On-Demand Treatment | PUPs -During Perioperative Management
Number analyzed (Participants) | 36 | 47 | 25
IU/kg | 87.1 [6.5 to 352.3] | 12.5 [2.4 to 176.8] | 606.4 [256.5 to 1951.0]

6. Secondary Outcome: In Vivo Incremental Recovery
Description: Change in factor VIII concentration from pre- to post-infusion at initial and termination study visits.
Time Frame: 30 minutes pre-infusion to 30 minutes post-infusion
Population: Participants who received pharmacokinetic rAHF-PFM infusions, did not develop inhibitors, and had assessments
Measure: Median (Full Range); unit: IU/dL per IU/kg
Groups:
- PUPs -Initial Visit: Incremental recovery at the Initial Study Visit
- PUPs -Termination Visit: Incremental recovery at the Termination Study Visit
Arm/Group | PUPs -Initial Visit | PUPs -Termination Visit
Number analyzed (Participants) | 4 | 12
IU/dL per IU/kg | 1.81 [0.74 to 1.92] | 1.71 [1.32 to 2.11]

7. Secondary Outcome: Assessment of Intra-operative Hemostasis
Description: Number of surgical procedures managed with rAHF-PFM and with surgeon's assessment of hemostasis based on a 4-point ordinal scale: Excellent: ≤ average predicted blood loss for matched procedures in healthy individuals Good: > average predicted blood loss, but ≤ maximal predicted blood loss for matched procedures in healthy individuals Fair: > maximal predicted blood loss for matched procedures in healthy individuals, and hemostasis was achieved None: uncontrolled hemostasis with proper dosing, necessitating a change in treatment regimen
Time Frame: Assessed at the time of discharge from recovery room
Population: Number of participants who underwent a surgical procedure with an intraoperative assessment of hemostatic efficacy
Measure: Number; unit: Procedures
Arm/Group | PUPs
Number analyzed (Participants) | 22
Procedures
  Excellent | 18
  Good | 4
  Not Applicable | 0
  Not Done | 0

8. Secondary Outcome: Assessment of Postoperative Hemostasis
Description: Number of surgical procedures managed with rAHF-PFM and with investigator's assessment of hemostasis based on a 4-point ordinal scale: Excellent: hemostasis was as good as or better than other licensed factor VIII products for matched procedure Good: hemostasis was probably as good as other licensed factor VIII products for matched procedure Fair: hemostasis was clearly < optimal for matched procedure, without need to change regimen None: bleeding from inadequate response with proper dosing, necessitating a change in regimen
Time Frame: Assessed at the time of discharge from hospital or clinic
Population: Number of participants who underwent a surgical procedure with a postoperative assessment of hemostatic efficacy
Measure: Number; unit: Procedures
Arm/Group | PUPs
Number analyzed (Participants) | 27
Procedures
  Excellent | 23
  Good | 2
  Not Applicable | 1
  Not Done | 1

9. Secondary Outcome: Assessment of Blood Loss During Surgical Procedures
Description: Percentage of actual intraoperative blood loss compared to preoperatively predicted average and maximal blood loss in hemostatically normal matched individuals (from institutional blood bank records)
Time Frame: Predicted volumes preoperatively estimated and actual volumes intraoperatively recorded
Population: Number of participants who underwent a surgical procedure with blood loss assessments
Measure: Median (Full Range); unit: Percentage Blood Loss
Arm/Group | PUPs
Number analyzed (Participants) | 27
Percentage Blood Loss
  Blood loss as percentage of predicted average | 50.0 [0.0 to 250]
  Blood loss as percentage of predicted maximal | 20.0 [0.0 to 100.0]

10. Secondary Outcome: Adverse Events Deemed Related to Treatment
Description: Percentage of participants who reported AEs deemed related to treatment with rAHF-PFM
Time Frame: Reported during the study period which was to be at least 75 exposure days or 3 years (whichever came first)
Population: Participants who received at least 1 infusion of rAHF-PFM
Measure: Number; unit: Percentage of Participants
Arm/Group | PUPs
Number analyzed (Participants) | 55
Percentage of Participants | 36.4

11. Secondary Outcome: Development of Antibodies to Heterologous Proteins
Description: Percentage of treated participants who developed antibodies to heterologous proteins (ie, Chinese Hamster Ovary Cell Protein, Murine IgG, or Recombinant Human VWF)
Time Frame: Assessed at baseline, throughout the duration of the study, which was to be at least 75 exposure days or 3 years (whichever came first), and at the termination visit.
Population: Participants who received at least 1 infusion of rAHF-PFM and had assessments of heterologous antibodies
Measure: Number; unit: Percentage of Participants
Arm/Group | PUPs
Number analyzed (Participants) | 55
Percentage of Participants
  Antibodies to Chinese Hamster Ovary Cell Protein | 0.00
  Antibodies to Murine IgG | 0.00
  Antibodies to Recombinant Human VWF (n=54) | 0.00

12. Post Hoc Outcome: Factor VIII Inhibitor Risk Factor: Genetic Risk Factor- Family History of Inhibitors
Description: Number of treated participants who developed an inhibitor
Time Frame: Duration of study which was to be at least 75 exposure days or 3 years (whichever came first)
Population: Immunogenicity Analysis Set- Participants who developed an inhibitor or who were inhibitor-free with ≥10 exposure days to rAHF-PFM
Measure: Number; unit: Participants
Arm/Group | PUPs - Did Not Develop Factor VIII Inhibitor | PUPs - Developed Factor VIII Inhibitor
Number analyzed (Participants) | 34 | 16
Participants
  Has Family History of Inhibitors | 6 | 8
  Unknown Family History of Inhibitors | 2 | 1
  No Family History of Inhibitors | 26 | 7
Statistical Analysis 1: Comparison: PUPs - Did Not Develop Factor VIII Inhibitor vs PUPs - Developed Factor VIII Inhibitor; Test type: Superiority or Other; Odds Ratio (OR) = 4.95, 95% CI [1.29 to 19.06]

13. Post Hoc Outcome: Factor VIII Inhibitor Risk Factor: Race
Description: Number of treated participants who developed an inhibitor
Time Frame: Duration of study which was to be at least 75 exposure days or 3 years (whichever came first)
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | PUPs - Did Not Develop Factor VIII Inhibitor | PUPs - Developed Factor VIII Inhibitor
Number analyzed (Participants) | 34 | 16
Participants
  Non-Caucasian | 8 | 9
  Caucasian | 26 | 7
Statistical Analysis 1: Comparison: PUPs - Did Not Develop Factor VIII Inhibitor vs PUPs - Developed Factor VIII Inhibitor; Test type: Superiority or Other; Odds Ratio (OR) = 4.18, 95% CI [1.18 to 14.82]

14. Post Hoc Outcome: Factor VIII Inhibitor Risk Factor: Number of Participants With Intensive Treatment and High Dose (≤20 Exposure Days (EDs))
Description: Immunogenicity Analysis Set- Participants with 5 consecutive study days of a mean infusion dose of FVIII >50 IU/kg within ≤20 EDs who developed an inhibitor
Time Frame: Duration of study which was to be at least 75 exposure days or 3 years (whichever came first)
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | PUPs - Did Not Develop Factor VIII Inhibitor | PUPs - Developed Factor VIII Inhibitor
Number analyzed (Participants) | 34 | 16
Participants
  Received intensive treatment & high dose | 4 | 6
  No intensive treatment & high dose | 30 | 10
Statistical Analysis 1: Comparison: PUPs - Did Not Develop Factor VIII Inhibitor vs PUPs - Developed Factor VIII Inhibitor; Test type: Superiority or Other; Odds Ratio (OR) = 4.50, 95% CI [1.05 to 19.25]

ADVERSE EVENTS:
Time Frame: Study period was to be at least 75 exposure days or 3 years (whichever came first)
Description: Median days on study was 498 (range: 82 to 1360) days. Median days of rAHF-PFM exposure was 76 (range: 1 to 414) exposure days.
Arm/Group | PUPs
Serious Adverse Events (participants affected / at risk) | 28/55
Other Adverse Events (participants affected / at risk) | 52/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PUPs (N=55)
Factor VIII inhibition (Blood and lymphatic system disorders) | 16 (16)
Coagulopathy (Blood and lymphatic system disorders) | 2 (3)
Mouth injury (Injury, poisoning and procedural complications) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Bronchitis (Infections and infestations) | 1 (1)
Catheter bacteraemia (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (3)
Catheter site haematoma (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PUPs (N=55)
Pyrexia (General disorders) | 39 (137)
Nasopharyngitis (Infections and infestations) | 28 (80)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (65)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 (54)
Diarrhea (Gastrointestinal disorders) | 20 (31)
Ear infection (Infections and infestations) | 20 (44)
Vomiting (Gastrointestinal disorders) | 17 (29)
Upper respiratory tract infection (Infections and infestations) | 16 (35)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 (48)
Rash (Skin and subcutaneous tissue disorders) | 13 (18)
Anaemia (Blood and lymphatic system disorders) | 10 (13)
Conjuctivitis (Eye disorders) | 9 (12)
Procedural pain (Injury, poisoning and procedural complications) | 9 (11)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 (8)
Otitis media (Infections and infestations) | 7 (13)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Hand-foot-and-mouth disease (Infections and infestations) | 5 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (8)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (5)
Bronchitis (Infections and infestations) | 4 (10)
Influenza (Infections and infestations) | 4 (8)
Pain (General disorders) | 4 (6)
Pharyngitis (Infections and infestations) | 4 (4)
Rhinitis (Infections and infestations) | 4 (14)
Varicella (Infections and infestations) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Croup infectious (Infections and infestations) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Gasteroenteritis (Infections and infestations) | 3 (3)
Mouth injury (Injury, poisoning and procedural complications) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3)
Viral infection (Infections and infestations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs vary per individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) 30 days prior to submission or communication. Baxter may request an additional delay of up to 90 days (e.g., to allow for intellectual property protection).